CLINICAL TRIAL: NCT02674035
Title: Plication of the Rectus Abdominis in Two Planes and in One Continuous Suture Plan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Luiz Jose Muaccad Gama (Other)
Responsible Party: Sponsor-Investigator, Luiz Jose Muaccad Gama, MD, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1175-1484
Record Dates: First submitted 2015-11-08; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Disorder of Abdomen
Keywords: Abdominoplasty; Sutures; Abdominal deformities; Plication; Monofilament nylon suture; Barbed suture
MeSH Terms: interventions — Abdominoplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Device: 2-0 monofilament nylon suture (Active Comparator): Plication of the anterior rectus sheath (correction of diastasis of the rectus abdominis muscles) was performed in two layers with Device 2-0 monofilament nylon suture (control group). Operative time was recorded. All patients underwent ultrasound examination preoperatively and at 3 weeks and 6 months postoperatively to monitor for diastasis recurrence. The force required to bring the anterior rectus sheath to the midline was measured at the supraumbilical and infraumbilical levels.
  Interventions: Procedure: Correction of diastasis of the rectus abdominis muscles
- Device: Single layer 2-0 monofilament (Active Comparator): Single layer with a Device 2-0 monofilament nylon suture (correction of diastasis of the rectus abdominis muscles) (group I). Operative time was recorded. All patients underwent ultrasound examination preoperatively and at 3 weeks and 6 months postoperatively to monitor for diastasis recurrence. The force required to bring the anterior rectus sheath to the midline was measured at the supraumbilical and infraumbilical levels.
  Interventions: Procedure: Correction of diastasis of the rectus abdominis muscles
- Device: Barbed suture Quill Nylon 1 (Active Comparator): Using a continuous Device Barbed suture Quill Nylon 1 (correction of diastasis of the rectus abdominis muscles) (group II). Operative time was recorded. All patients underwent ultrasound examination preoperatively and at 3 weeks and 6 months postoperatively to monitor for diastasis recurrence. The force required to bring the anterior rectus sheath to the midline was measured at the supraumbilical and infraumbilical levels.
  Interventions: Procedure: Correction of diastasis of the rectus abdominis muscles

INTERVENTIONS:
Procedure: Correction of diastasis of the rectus abdominis muscles — Thirty women with similar abdominal deformities, who had had at least one pregnancy, were randomized into three groups to undergo abdominoplasty. Plication of the anterior rectus sheath was performed in two layers with 2-0 monofilament nylon suture (control group) or in a single layer with either a continuous 2-0 monofilament nylon suture (group I) or using a continuous barbed suture (group II). Operative time was recorded. All patients underwent ultrasound examination preoperatively and at 3 weeks and 6 months postoperatively to monitor for diastasis recurrence. The force required to bring the anterior rectus sheath to the midline was measured at the supraumbilical and infraumbilical levels.
  Other Names: Abdominoplasty

SUMMARY:
Thirty women with similar abdominal deformities, who had had at least one pregnancy, were randomized into three groups to undergo abdominoplasty. Plication of the anterior rectus sheath was performed in two layers with 2-0 monofilament nylon suture (control group) or in a single layer with either a continuous 2-0 monofilament nylon suture (group I) or using a continuous barbed suture (group II). Operative time was recorded. All patients underwent ultrasound examination preoperatively and at 3 weeks and 6 months postoperatively to monitor for diastasis recurrence. The force required to bring the anterior rectus sheath to the midline was measured at the supraumbilical and infraumbilical levels.

DETAILED DESCRIPTION:
Inclusion criteria were female gender; 25 to 50 years of age; history of at least one pregnancy; body mass index (BMI) between 18 and 30 kg/m2; desire to undergo abdominoplasty as a single procedure without receiving liposuction or other cosmetic surgeries; deformities of the skin and subcutaneous tissues in the abdominal region; and musculoaponeurotic defect.

Non-inclusion criteria were smoking habit; abdominal wall scar (except for a Pfannenstiel scar related to a Cesarean section); abdominal wall hérnias; history of deep-vein thrombosis; chronic obstructive pulmonary disease; câncer; hypertension; diabetes or other chronic systemic diseases; and use of corticosteroids. Patients lost to follow-up and those who did not undergo ultrasound examination were excluded from the study.

Primary outcome: Get a technique that provides a safe correction with lasting results and in every segment of time.

Secondary clinical outcome: confirms the plication of a single layer as positive in women patients at two years of surgery compared to two planes.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age: 25 to 50 years of age
* History of at least one pregnancy
* Body mass index (BMI) between 18 and 30 kg/m2
* Desire to undergo abdominoplasty as a single procedure without receiving liposuction or other cosmetic surgeries
* Deformities of the skin and subcutaneous tissues in the abdominal region
* Musculoaponeurotic defect

Exclusion Criteria:

* Smoking habit;
* Abdominal wall scar (except for a Pfannenstiel scar related to a Cesarean section);
* Abdominal wall hérnias;
* History of deep-vein thrombosis;
* Chronic obstructive pulmonary disease;
* Câncer;
* Hypertension;
* Diabetes or other chronic systemic diseases;
* Use of corticosteroids.
* Patients lost to follow-up and those who did not undergo ultrasound examination were excluded from the study

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Correction of diastasis of the rectus abdominis muscles | Compare from the baseline the efficacy and time required to correct the diastasis at 3 weeks
  Get a technique that provides a safe abdominoplasty correction with lasting results and in every segment of time.

SECONDARY OUTCOMES:
Follow-up of diastasis of the rectus abdominis muscles | At six months
  Confirms the plication of a single layer abdominoplasty as positive in women patients at six months of surgery compared to two planes.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz José Muaccad Gama, MD, Principal Investigator — Universidade Federal de São Paulo - UNIFESP
Locations (1):
- Fábio Xerfan Nahas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No